CLINICAL TRIAL: NCT04884282
Title: A Multicenter, Phase II, Open Label, Randomized Trial Evaluating the Efficacy of Tedopi Plus Docetaxel or Tedopi Plus Nivolumab as Second-line Therapy in Metastatic Non-small-cell Lung Cancer Progressing After First-line Chemo-immunotherapy (Combi-TED)
Brief Title: Efficacy of Tedopi Plus Docetaxel or Tedopi Plus Nivolumab as Second-line Therapy in Metastatic Non-small-cell Lung Cancer Progressing After First-line Chemo-immunotherapy (Combi-TED)
Acronym: COMBI-TED
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBI-TED
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A - tedopi + docetaxel (Experimental): Tedopi every 3 weeks plus docetaxel every 3 weeks only for 6 cycles, then maintenance with Tedopi alone every 6 weeks until the end of year 1, then every 12 weeks until disease progression, unacceptable toxicity or patient refusal.
  Interventions: Drug: Tedopi; Drug: Docetaxel
- Arm B - tedopi + nivolumab (Experimental): Tedopi every 3 weeks plus nivolumab 360 mg every 3 weeks for 6 cycles, then maintenance nivolumab 360 mg every 3 weeks plus Tedopi every 6 weeks until the end of year 1, then every 12 weeks until disease progression, unacceptable toxicity or patient refusal
  Interventions: Drug: Tedopi; Drug: Nivolumab
- Arm C - docetaxel (Other): Docetaxel every 3 weeks until disease progression, unacceptable toxicity, patient refusal, or for a maximum of 6 cycles (whichever comes first).
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Tedopi — TEDOPI is a T-specific immunotherapy was designed to induce cytotoxic T-lymphocytes against five five tumor associated antigens (ie CEA, p53, HER-2/neu, MAGE2 and MAGE3)
  Arms: Arm A - tedopi + docetaxel; Arm B - tedopi + nivolumab
Drug: Nivolumab — Nivolumab is a soluble protein consisting of 4 polypeptide chains, which include 2 identical heavy chains and 2 identical light chains. Nivolumab is produced from cell culture using a CHO cell line.
  Arms: Arm B - tedopi + nivolumab
Drug: Docetaxel — Docetaxel is a cytotoxic microtubule inhibiting antineoplastic agent in the taxane class. Docetaxel monotherapy is indicated for locally advanced or metastatic NSCLC after failure of prior platinum- based chemotherapy.
  Arms: Arm A - tedopi + docetaxel; Arm C - docetaxel

SUMMARY:
This is a phase II, non-comparative, randomized study assessing combination of Tedopi with docetaxel or with nivolumab in NSCLC patients failing after first- line chemoimmunotherapy. In this non-comparative study, the standard arm (arm C) will serve as a calibration arm. All NSCLC patients candidate for second- line therapy are considered eligible for the study if they are HLA-A2+ and if they progressed after at least 4 cycles of previous first-line chemo-immunotherapy. After evaluation of all inclusion and exclusion criteria and after informed consent signature, all eligible patients will be treated with Tedopi plus docetaxel (arm A) or Tedopi plus nivolumab (arm B) or docetaxel as single agent (arm C- standard arm). Docetaxel therapy will be given until disease progression, unacceptable toxicity or patient refusal, and up to maximum 6 cycles. Tedopi or nivolumab will be given until disease progression, unacceptable toxicity or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients willing and able to give written informed consent;
2. Histological or cytological confirmed diagnosis of HLA-A2+ NSCLC with no evidence of EGFR mutations or ALK or ROS1 rearrangement;
3. Evidence of disease progression at the end of at least 4 cycles of chemo-immunotherapy or 2 cycles of chemo-immunotherapy followed by 2 cycles of immunotherapy (CheckMate9LA regimen) and eligible for treatment with docetaxel. This criterion implies that patients with immunotherapy primary resistance are excluded;
4. Patients must have experienced progressive disease (PD), either during or within 3 months of discontinuing treatment with anti-PD-(L)1-based therapy, occurring after previous clear benefit (any complete -CR- or partial response -PR), or after previous stable disease (SD);
5. Performance status 0-1 (ECOG);
6. Patient compliance to trial procedures;
7. Age ≥ 18 years;
8. Adequate BM function (ANC ≥ 1.5x109/L, Platelets ≥ 100x109/L, HgB > 9g/dl);
9. Adequate liver function (bilirubin < G2, transaminases no more than 3xULN/<5xULN in present of liver metastases);
10. Normal level of creatinine;
11. Female patient: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [complete abstinence, intrauterine contraceptive device (IUD), birth control pills, or barrier device] until 5 months after end of treatment.

    or Male patient: should practice complete abstinence or if sexually active with WOCBP must use any contraceptive method with failure rate less than 1%/year and they should not donate semen as follows: in arm A and C until 6 months since the last dose of docetaxel; in arm B until 3 months since last dose of tedopi.
12. Prior palliative radiotherapy to non-CNS lesions must have been completed at least 2 weeks prior to treatment. Subjects with symptomatic tumor lesions that may require palliative radiotherapy within 4 weeks of first treatment are strongly encouraged to receive palliative radiotherapy prior to treatment. Patients are eligible if CNS metastases are adequately treated and patients are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to randomization;
13. Patients must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) for at least 2 weeks prior to randomization.

Exclusion Criteria:

1. Patient positive for actionable EGFR mutations or ALK or ROS1 rearrangement;
2. No previous chemoimmunotherapy for metastatic disease or evidence of disease progression during the first 4 cycles of chemoimmunotherapy (primary resistance). Patients with adjuvant resistance (documented loco-regionally and/or systemic relapse of their disease occurring <6 months after the last dose of anti-PD-(L)1-based systemic adjuvant therapy) are excluded;
3. Patients with intervening systemic therapy following prior anti-PD-(L)1-based therapy;
4. Symptomatic brain metastases. Asymptomatic brain metastases are allowed if not requiring corticosteroids use at a dose >10mg daily prednisone (or equivalent);
5. Diagnosis of any other malignancy during the last 3 years, except for in situ carcinoma of cervix uteri and cutaneous squamous cell carcinoma or other local tumors considered cured;
6. Pregnancy or lactating;
7. Patients with an active, known or suspected autoimmune disease. Patients with type I diabetes mellitus; hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll;
8. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease;
9. Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection;
10. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year Survival Rate | 1 year
  1-year Survival Rate

CONTACTS AND LOCATIONS:
Locations (23):
- France (4):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Cholet, Cholet
  - GHR Mulhouse Sud Alsace - Hôpital Emile Muller, Mulhouse
  - Nouvel Hôpital Civil - Hopitaux Universitaires de Strasbourg, Strasbourg
- Italy (13):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forlì
  - AO Busto Arstizio PO Saronno, Saronno, Varese
  - Ospedale Mater Salutis Legnago, Legnago, Verona
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Ospedale San Paolo, Civitavecchia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AOOR Papardo-Piemonte, Messina
  - AOU "Maggiore della Carità", Novara
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera di Perugia, Perugia
  - IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - ASST Sette Laghi, Varese
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Clinica Mi Tres Torres - UOMI Cancer Center, Barcelona
  - Vall d'Hebron Universitary Hospital, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Universitario Regional de Málaga - Hospital Civil, Málaga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Landi L, Delmonte A, Bonetti A, Pasello G, Metro G, Mazzoni F, Borra G, Giannarelli D, Andrikou K, Mangiola D, Gori S, D'Andrea MR, Minuti G, Resuli B, Laudisi A, Vidiri A, Conti L, Cappuzzo F. Combi-TED: a new trial testing Tedopi(R) with docetaxel or nivolumab in metastatic non-small-cell lung cancer progressing after first line. Future Oncol. 2022 Dec;18(40):4457-4464. doi: 10.2217/fon-2022-0913. Epub 2023 Mar 22. PMID 36946237